CLINICAL TRIAL: NCT06750874
Title: Feasibility and Acceptability of a Single-session Perioperative Acceptance and Commitment Therapy (ACT) Workshop for Preventing Chronic Postsurgical Pain: a Single-arm, Non-randomized Pilot Trial
Brief Title: Perioperative ACT for Preventing CPSP: a Single-arm Non-randomized Pilot Trial
Acronym: PREPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samantha Meints (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor-Investigator, Samantha Meints, Assistant Professor, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020A003336; K23AR077088 (NIH)
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Back Pain; Spinal Stenosis; Spondylosis; Spondylolisthesis; Back Injury
Keywords: acceptance and commitment therapy; chronic postsurgical pain; ACT
MeSH Terms: conditions — Back Pain; Spinal Stenosis; Spondylosis; Spondylolisthesis; Back Injuries; Pain, Postoperative | interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Intervention Model Description: Non-randomized, non-controlled pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Perioperative Acceptance and Commitment Therapy Workshop (Experimental): Participants assigned to this arm will complete a 1-day ACT workshop followed by a telephone booster after surgery
  Interventions: Behavioral: Acceptance and Commitment Therapy

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy — One day workshop + telephone booster

SUMMARY:
The present study aims to adapt and modify a brief perioperative Acceptance and Commitment Therapy (ACT) intervention aimed at preventing the transition to Chronic Post-Surgical Pain (CPSP) and reducing long-term opioid use. Investigators will assess the acceptability, feasibility, and preliminary efficacy of the intervention via a non-randomized, non-controlled pilot trial.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to undergo fusion, discectomy, vertebroplasty, kyphoplasty, or foraminotomy
* age 22 and older
* able to communicate fluently in English

Exclusion Criteria:

* inability to complete study procedures due to delirium, dementia, psychosis, or other cognitive impairment
* have a history of severe neurologic movement disorder
* are pregnant or intent to become pregnant during study
* have undergone previous spinal surgery
* have spinal deformity, pseudarthrosis, trauma, infection, or tumor as primary indication for surgery
* have undergone Acceptance and Commitment Therapy in last 2 years

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Treatment helpfulness (THQ) | Immediately following the ACT workshop
  Item assesses the perceived helpfulness of the ACT workshop and is rated from -5 (extremely harmful) to 5 (extremely helpful).

SECONDARY OUTCOMES:
Treatment Helpfulness (THQ) | 1 month post-op
  Item assesses the perceived helpfulness of the ACT workshop and is rated from -5 (extremely harmful) to 5 (extremely helpful).
Treatment Credibility | immediately following ACT workshop
  Credibility and Expectancy Questionnaire (CEQ); 3 items are rated to indicate the logic, success, and confidence in the treatment. Scores are summed with a range from 3-27 where higher scores indicating greater treatment credibility
Treatment Expectancy | immediately following ACT workshop
  Credibility and Expectancy Questionnaire (CEQ); 3 items are used to assess the likelihood of the success of the therapy to reduce pain and improve function. Scores are summed with a range from 0-29 where higher scores indicate greater expectancy for beneficial treatment outcomes
Pain Interference | 1 month post-op
  Assesses how much a person's pain impacts their daily activities, including general activity, mood, walking, work, relationships with others, enjoyment of life, and sleep, with higher scores indicating greater interference with daily functioning due to pain. Each of the seven domains is rated on a scale from 0 (no interference) to 10 (complete interference), and the average score across these domains represents the overall pain interference level.
Pain Interference | 3 months post-op
  The Brief Pain Inventory assesses how much a person's pain impacts their daily activities, including general activity, mood, walking, work, relationships with others, enjoyment of life, and sleep, with higher scores indicating greater interference with daily functioning due to pain. Each of the seven domains is rated on a scale from 0 (no interference) to 10 (complete interference), and the average score across these domains represents the overall pain interference level.
Pain Interference | 6 months post-op
  The Brief Pain Inventory assesses how much a person's pain impacts their daily activities, including general activity, mood, walking, work, relationships with others, enjoyment of life, and sleep, with higher scores indicating greater interference with daily functioning due to pain. Each of the seven domains is rated on a scale from 0 (no interference) to 10 (complete interference), and the average score across these domains represents the overall pain interference level.
Pain Severity | 1 month post-op
  The Brief Pain Inventory (BPI) measures pain severity by asking patients to rate their "worst pain" on a scale from 0 to 10, where a higher score indicates greater pain intensity
Pain Severity | 3 months post-op
  The Brief Pain Inventory (BPI) measures pain severity by asking patients to rate their "worst pain" on a scale from 0 to 10, where a higher score indicates greater pain intensity
Pain Severity | 6 months post-op
  The Brief Pain Inventory (BPI) measures pain severity by asking patients to rate their "worst pain" on a scale from 0 to 10, where a higher score indicates greater pain intensity

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Upon publication of the primary study manuscript
Access Criteria: Reasonable requests from IPD will be reviewed and granted by the study PI.